CLINICAL TRIAL: NCT02765347
Title: The Effects of Metformin on Glycemic Control and Insulin Sensitivity in Adolescents With T1DM: A Randomized, Cross-over, Prospective Study
Brief Title: The Effects of Metformin on Glycemic Control and Insulin Sensitivity in Adolescents With T1DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wen Xu, Associated Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016-T1DM
Record Dates: First submitted 2016-02-14; First posted 2016-05-06 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Metformin; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin and Insulin (Other): MDI or CSII plus metformin (initially starting dosage with 0.5g qd, then gradually increasing to 0.5g bid or tid) for 24 weeks
  Interventions: Drug: Metformin
- Insulin (Other): Accept insulin for 24 weeks
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Metformin — For arm 1, accept MDI or CSII plus metformin (initially starting dosage with 0.5g qd, then gradually increasing to 0.5g tid) for 24 weeks.
  Other Names: Glucophage
  Arms: Metformin and Insulin
Drug: Insulin — For arm 2, just accept insulin for 24 weeks
  Other Names: CSII or MDI
  Arms: Insulin

SUMMARY:
The investigators intends to carry out a randomized, cross-over, prospective study which will last 48 weeks in youth with T1DM followed up by the center. The purpose is to observe the effects of metformin on glycemic control and insulin sensitivity in adolescents with T1DM based on insulin therapy by using 72h CGMS and hyperinsulinemic euglycemic clamps.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes mellitus;
2. Age≥12 yr;
3. Tanner sexual maturation rating 2-5;
4. HbA1c levels: 7.5%-10%;
5. MDI or CSII ≥6 months;
6. Insulin dose ≥ 0.8U/kg before the enrollment，and the dosage is stable at least >1 month（dosage change<10%）.

Exclusion Criteria:

1. Serious acute and chronic complications associated with diabetes;
2. Repeated and serious hypoglycemia episodes repeatedly;
3. Hepatic function damage (ALT≥2.5 times higher than the upper limit of the normal accepted range);
4. Moderate to advanced renal impairment (calculated according to MDRD equation: eGFR<60ml/min/1.73m2);
5. Clinically significant heart attacks: myocardial infarction, arrhythmia，II-III°AVB，unstable angina，decompensated HF（NYHA III~IV;
6. Female patients who have a sex life and are not willing to use contraceptive methods;
7. Pregnancy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
HbA1c | half one year

CONTACTS AND LOCATIONS:
Overall Officials: Wen Xu, Principal Investigator — Associated professor
Locations (1):
- The Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided